CLINICAL TRIAL: NCT00479856
Title: An Open-label, Multi-centre Study of Lapatinib in Combinationwith Chemotherapy in Patients With ErbB2 Overexpressing Breastcancer After Trastuzumab Failure in the Neoadjuvant or Adjuvantsetting.
Brief Title: Lapatinib In Combination With Chemotherapy In Subjects With Relapsed Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to difficulty in identifying eligible subjects
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF108916
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Results first posted 2010-06-02 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2011-06

CONDITIONS: Relapsed Breast Cancer; Neoplasms, Breast
Keywords: ErbB1; ErbB2; GW572016; lapatinib; Relapsed breast cancer; dual tyrosine kinase inhibitor; MBC; EGFR; Her-2/neu; FISH amplification
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Capecitabine; Docetaxel; 130-nm albumin-bound paclitaxel

ARMS (1):
- Lapatinib plus Chemotherapy (Experimental): Lapatinib is administered in combination with one of the following chemotherapies based on the discretion of the investigator : capecitabine, docetaxel or nab-paclitaxel.
  Interventions: Drug: Lapatinib; Drug: Capecitabine; Drug: Docetaxel; Drug: nab-Paclitaxel

INTERVENTIONS:
Drug: Lapatinib — Small molecule tyrosine kinase inhibitor
Drug: Capecitabine — Chemotherapy
Drug: Docetaxel — Chemotherapy
Drug: nab-Paclitaxel — Chemotherapy

SUMMARY:
This study will evaluate the safety and efficacy of lapatinib in combination with chemotherapy (capecitabine, docetaxel, nab-paclitaxel) in subjects with ErbB2-overexpressing breast cancer whose disease has progressed during or within 12 months after completion of trastuzumab-containing therapy in the neoadjuvant or adjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Histologically/cytologically confirmed breast cancer;

If the disease is restricted to a solitary lesion, the neoplastic nature of the lesion must be confirmed by cytology or histology.

* Measurable lesion(s) according to RECIST (Response Evaluation Criteria in Solid Tumors) [Therasse, 2000].
* Documented amplification of the ErbB2 gene by fluorescence in situ hybridization (FISH) or documented overexpression of the ErbB2 protein by 3+ IHC in primary or metastatic tumor tissue.
* Subjects must have relapsed breast cancer where the disease progressed during or ≤ 12 months after completion of trastuzumab-containing therapy in the neoadjuvant or adjuvant setting.

Note: Progression is defined using RECIST criteria, that is, either the appearance of new lesions or a >=20% increase in the sum of longest diameter (LD).

* Subjects must not have received prior anti-cancer therapy for metastatic breast cancer (MBC). Subjects who received prior antihormonal agents combined with trastuzumab for the treatment of disease which first presented as ER positive MBC and recurred while receiving trastuzumab or ≤ 3 months after completing this therapy are eligible.
* Subjects with stable central nervous system (CNS) metastases as confirmed by computerized tomography (CT)/magnetic resonance imaging (MRI) are allowed. Treatment with prophylactic anticonvulsants is permitted, unless listed within the Prohibited Medications.
* Subjects must have a baseline cardiac ejection fraction (LVEF) ³50% measured by echocardiogram (ECHO) (or multigated acquisition (MUGA) scan if an ECHO cannot be performed). The same modality used at baseline must be used for repeat assessment throughout study. Only subjects with controlled or asymptomatic angina or arrhythmias are eligible.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 2.
* Subjects must have archived tumor tissue from the initial diagnosis available for analysis. If tissue from the initial diagnosis is not available, then tissue must be obtained from a recurrent or metastatic site prior to initiating study treatment.
* Female ≥18 years.
* Subject must have adequate organ function as defined in Table 1.
* Table 1: Baseline Laboratory Values for Adequate Organ Function.

SYSTEM

Hematologic:

Absolute neutrophil count: ≥1.5 X 10^9/L

Hemoglobin: ≥9 g/dL

Platelets: ≥ 75 X 10^9/L

Hepatic:

AST, ALT and Alkaline phosphatase: ≤ 2.5 X ULN

Unless concomitant docetaxel, then ≤ 1.5 x ULN for AST and ALT, with AP ≤ 2.5 x ULN

Unless documented liver metastasis, then ≤ 5 x ULN

Serum bilirubin: ≤ 2.0 X ULN

Albumin: ≥ 2.5 g/dL

Renal:

Serum Creatinine: ≤ 1.5 mg/dL

* OR - Calculate Creatinine Clearance: ≥ 40 mL/min

  1. Calculated by the Cockcroft and Gault Method [Cockcroft , 1976].

Exclusion Criteria:

* Pregnant or lactating females.
* Women of childbearing potential who do not practice approved contraceptive methods (for example, intrauterine device [IUD], birth control pills, or barrier device) beginning 2 weeks before the first dose of investigational product and for 28 days after the final dose of investigational product.
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Concurrent therapy given to treat cancer (chemotherapy, radiation therapy, immunotherapy, biologic therapy, anti-hormonal therapy) while taking study medication.
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment.
* Malabsorption syndrome or resection of the stomach or small bowel significantly affecting gastrointestinal function.
* Have current active haptic or biliary disease (with excpetion of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
* Concurrent disease or condition that, in the opinion of the physician, would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety (for example, uncontrolled infection, or any psychiatric condition prohibiting understanding or rendering of informed consent).
* Concurrent treatment with an investigational agent or participation in another clinical trial involving investigational agents for anti-cancer therapy.
* Bisphosphonates may not be initiated after the first dose of study medication.
* Considered by the Investigator to have a life expectancy less than 3 months.
* Not able to swallow or retain oral medication.
* The subject with a known unmanageable hypersensitivity reaction or idiosyncrasy to drugs chemically related to lapatinib or excipients and those related to capecitabine, docetaxel, nab paclitaxel or their excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (28):
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Highland, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Zion, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Tupelo, Mississippi
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Sumter, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib + Chemotherapy: 1250 milligrams (mg) Lapatinib taken once daily on a continuous basis plus one of the following chemotherapies:
  (1) 1000 mg/square meters (m2) Capecitabine taken twice a day on Days 1-14 every 21 days; (2) 75 mg/m2 Docetaxel administered as a single infusion once every 21 days; or (3) 100 mg/m2 nab-Paclitaxel administered as a single infusion once every 7 days for 21 days, followed by 7 days of rest in a 28-day cycle
Period: Overall Study
Arm/Group | Lapatinib + Chemotherapy
Started | 9
Completed | 6
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib + Chemotherapy
Number analyzed (Participants) | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 61.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 7
  African American/African Heritage | 1
  American Indian or Alaska Native | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumor Response
Description: Overall tumor response is defined as the percentage of participants with a confirmed complete or partial tumor response per Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is defined as the disappearance of all target lesions. CR could only be declared if all target and non-target lesions had disappeared. Partial response (PR) is defined as a decrease of 30% or greater in the sum of the longest diameter of target lesions.
Time Frame: from start of treatment and every 6 weeks (wks) until Wk 12, then every 12 wks thereafter through the end of treatment (~95 wks; dependent on when participant discontinued study therapy due to disease progression, death, adverse event, of other reason)
Population: All Treated Subjects (ATS) Population: all participants who received at least one dose of study treatment
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib + Chemotherapy
Number analyzed (Participants) | 9
percentage of participants | 33.3
Statistical Analysis 1: Comparison: Lapatinib + Chemotherapy; Test type: Superiority or Other; percentage of participants = 33.3, 95% CI [7.5 to 70.1]

2. Secondary Outcome: Clinical Benefit (CB)
Description: CB is defined as the percentage of participants (par.) with either a confirmed CR or PR or stable disease (SD) for at least 24 weeks. SD is defined as small changes that do not meet criteria for CR, PR, or Progressive Disease (defined as at least a 20% increase in the sum of the longest diameter of target lesions).
Time Frame: from start of treatment and every 6 weeks (wks) until Wk 12, then every 12 wks thereafter through the end of treatment (~95 weeks; dependent on when participant discontinued study therapy due to disease progression, death, adverse event, or other reason)
Population: Due to the low incidence of relapse and hence the difficulty in identifying eligible par., the study was terminated with only 9 out of the 45 planned par. enrolled. As there were too few par. to derive statistically meaningful conclusions, only the primary endpoint was evaluated.
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib + Chemotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response
Description: For the subset of participants with a confirmed CR or PR, duration of response was measured as the time from first documented evidence of CR or PR until the first documented sign of disease progression or death.
Time Frame: time from first documented evidence of CR or PR until the first documented sign of disease progression or death (approximately 95 weeks)
Population: Due to the low incidence of relapse and hence the difficulty in identifying eligible participants, the study was terminated with only 9 out of the 45 planned participants enrolled. As there were too few participants to derive statistically meaningful conclusions, only the primary endpoint was evaluated.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib + Chemotherapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time from the start of treatment until the first documented evidence of PR or CR (whichever status was recorded first). When tumor response was confirmed at a repeat assessment, the TTR was taken to be the first time that the response was observed.
Time Frame: start of treatment until first documented evidence of CR or PR (approximately 95 weeks)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib + Chemotherapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-free Survival
Description: The time from the start of treatment until the earliest date of disease progression or death due to any cause was measured.
Time Frame: from start of treatment and every 6 weeks (wks) until Wk 12, then every 12 wks thereafter through the end of treatment (~95 weeks); dependent on when participant discontinued study therapy due to disease progression, death, adverse event, or other reason)
Population: Due to the low incidence of relapse and hence the difficulty in identifying eligible participants, the study was terminated with only 9 out of the 45 planned participants enrolled. As there were too few participants to derive statistically meaningful conclusions, only the primary endpoint of overall response rate was evaluated.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib + Chemotherapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With the Indicated Serious Adverse Events and Adverse Events
Description: Qualitative and quantitative toxicities associated with the combination of capecitabine, docetaxel, or nab-paclitaxel and lapatinib were measured. Data are presented as serious adverse events (SAEs) and adverse events (AEs). See the SAE/AE section of the results record for data.
Time Frame: Baseline through End of Treatment, or discontinuation of study therapy (approximately 95 weeks); from the first dose of lapatinib until 5 days after the last dose of lapatinib
Measure: Number; unit: participants
Arm/Group | Lapatinib + Chemotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Time from the first dose of lapatinib until 5 days after the last dose of lapatinib.
Arm/Group | Lapatinib + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Chemotherapy (N=9)
Small intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib + Chemotherapy (N=9)
Diarrhoea (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 7
Nausea (Gastrointestinal disorders) | 6
Palmar plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Dyspesia (Gastrointestinal disorders) | 2
Mucosal inflammation (General disorders) | 2
Urinary tract infection (Infections and infestations) | 2
Aspartatate aminotransferase increased (Investigations) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Feeling cold (General disorders) | 1
Local swelling (General disorders) | 1
Pain (General disorders) | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Paronychia (Infections and infestations) | 1
Periorbital cellulitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Weight decreased (Investigations) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Conjunctivitis (Eye disorders) | 1
Insomnia (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.